CLINICAL TRIAL: NCT05282238
Title: Quantification of Inspiratory Effort Through Nasal Pressure in Patients Undergoing Weaning From Invasive Mechanical Ventilation and Correlation With Clinical Outcomes
Acronym: NAIVE
Status: Not yet recruiting | Type: Observational
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Roberto Tonelli, Principal Investigator, University of Modena and Reggio Emilia
Other Study IDs: UModenaReggio15
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Respiratory Failure
Keywords: Weaning Failure; Inspiratory Effort; Nasal Pressure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Nasal pressure assessment — Once the patient is enrolled nasal pressure will be measured through a dedicated pressure line located at the nostril entrance and connected to a dedicated pressure transducer (OptiVentTM, SIDAM, Mirandola, Italy). Measured nasal pressure will be the result of the variation between inspiratory and expiratory pressure (DeltaPnose). The measurement of DeltaPnose will be obtained considering the average of 3 values registered during 3 breath after at least 3 minutes of stable and constant respiratory pattern. Pnose values will be measured before extubation (T0) and 30 minutes (T1), 2 hours (T2), 4 hours (T3), 12 hours (T4) , 24 hours (T5) and 48 hours (T6) after extubation.

SUMMARY:
Weaning from invasive mechanical ventilation (MV) constitutes a fundamental procedure in intensive care, covering up to 50% of time spent on ventilation (1). Endotracheal tube (ETT) removal might be an important but delicate step in intensive care setting. Failure and subsequent need for re-intubation can occur in up to 20% of cases leading to a significant increase in mortality rates (24%), longer hospital stay and prolonged need for ventilation. Comorbidities such as obesity, COPD and cardiac related diseases might further increase this risk reaching up to 60% of failure in extubation. In this scenario, accurate predictors of weaning failure are far welcomed. The recurrence of respiratory failure after extubation might considerably raise rates of failure, probably due to increased work of breathing in patients after ETT removal. Most recent guidelines on the use of non-invasive ventilation (NIV) suggest using NIV after ETT removal in subjects with high risk of failure. NIV could contribute to reduce work of breathing hence preventing the onset of respiratory failure after extubation. Therefore, measuring inspiratory effort and its variation in weaned patients might help in identifying patients with significant risk of failing extubation. Esophageal pressure swings (DeltaPES) can be measured through a nasogastric tube with a pressure transducer located in the inferior part of the esophagus. DeltaPES is an extremely precise and accurate method to quantify inspiratory effort, however its use in daily clinical practice is limited due to the invasive nature of the maneuver, elevated costs and need for considerable clinical training of operators. Physiological studies have shown a correlation between nasal pressure measured at nostril entrance and esophageal pressure (which in turn is a measure of respiratory effort .

Therefore, measuring nasal pressure could represent a method to quantify inspiratory effort non-invasively, proving to be useful in daily clinical practice.

ELIGIBILITY:
Inclusion Criteria:

- candidates for endotracheal tube removal.

Exclusion Criteria:

* Age under 18
* Pregnancy
* Patient unable or unwilling to sign informed consent
* Neuromuscular diseases
* Patient with compromised neurological state (Glasgow Coma Scale (GCS) under 14/15)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients will be enrolled among patients admitted in Intensive Care Unit of Azienda Ospedaliero-Universitaria Policlinico di Modena undergoing endotracheal intubation and mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 175 (Estimated)
Dates: Start 2027-05-01 (Estimated); Primary Completion 2030-05-01 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Weaning failure | 48 hours
  Weaning failure will be defined by need for re-intubation

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero Universitaria Policlinico di Modena, Modena, Italy

IPD SHARING:
Plan to Share IPD: No